CLINICAL TRIAL: NCT05409924
Title: The ATTRACTIVE 1 Trial - a First-in-human Phase I, Dose Escalating, Double-blind, Placebo-controlled, Single and Multiple Dose Trial of ATR-258 in Healthy Participants and Participants With Type 2 Diabetes Mellitus
Brief Title: First-in-human Single and Multiple Dose Trial of ATR-258
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atrogi AB (Industry)
Collaborators: Key2Compliance (Industry); CRS Clinical Research Services Mannheim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ATR-258-study-1
Record Dates: First submitted 2022-05-13; First posted 2022-06-08 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase A (Experimental): ATR-258 Single Ascending Dose or placebo
  Interventions: Drug: ATR-258
- Phase B (Experimental): ATR-258 Multiple Ascending Dose or placebo
  Interventions: Drug: ATR-258
- Phase C (Experimental): ATR-258 Repeated dosing or placebo
  Interventions: Drug: ATR-258

INTERVENTIONS:
Drug: ATR-258 — Single Ascending Dose
  Other Names: Placebo
  Arms: Phase A
Drug: ATR-258 — Multiple Ascending Dose
  Other Names: Placebo
  Arms: Phase B
Drug: ATR-258 — Repeat Dose
  Other Names: Placebo
  Arms: Phase C

SUMMARY:
This is a single-site, randomized, double-blinded, placebo-controlled, First-in-Human trial, conducted in 3 parts.

ELIGIBILITY:
Inclusion Criteria Phase A and B:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Body mass index (BMI) within the range 18.5 - 29.9 kg/m2 (inclusive) at screening.
* Male

Inclusion Criteria Phase C:

* Participant must be 30 to 75 years of age inclusive, at the time of signing the informed consent.
* BMI within the range 25.0 to 45.0 kg/m2 and body weight from 80 to 160 kg (inclusive) at screening.
* Male

Exclusion Criteria Phase C:

* Type 1 diabetes mellitus (T1DM) or ketosis-prone T2D based on diagnosis

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Safety analyses after single dose of ATR-258 | maximum 7 days post dosing
  Safety analyses will be performed based in incidence of TEAEs after single dose of ATR-258
Safety analyses after multiple doses of ATR-258 | maximum 56 days post dosing
  Safety analyses will be performed based in incidence of TEAEs after multiple doses of ATR-258

SECONDARY OUTCOMES:
PK analyses will be performed after PK of ATR-258 single dose | maximum 7 days post dosing
  PK analyses will be performed based on AUC0-inf of ATR-258 in plasma
PK analyses will be performed after PK of ATR-258 single dose | maximum 7 days post dosing
  PK analyses will be performed based on AUC0-tz of ATR-258 in plasma
PK analyses will be performed after PK of ATR-258 single dose | maximum 7 days post dosing
  PK analyses will be performed based on Cmax of ATR-258 in plasma
PK analyses will be performed after PK of ATR-258 multiple dose | maximum 56 days post dosing
  PK analyses will be performed based on AUCtau of ATR-258 in plasma
PK analyses will be performed after PK of ATR-258 multiple dose | maximum 56 days post dosing
  PK analyses will be performed based on AUC0-tz,MD of ATR-258 in plasma
PK analyses will be performed after PK of ATR-258 multiple dose | maximum 56 days post dosing
  PK analyses will be performed based on Cmax,MD of ATR-258 in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services, Mannheim, Germany

REFERENCES:
- See also: Related Info — https://atrogi.com/